CLINICAL TRIAL: NCT02435615
Title: Diagnosing Dengue: Evaluating the Utility of Oral Fluid for Dengue Diagnosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: An unexpected Zika outbreak prevented recruitment of study participants. The samples collected were subsequently destroyed and not analyzed.
Sponsor: University of Miami (Other)
Collaborators: Instituto Nacional de la Diabetes (Unknown); Hospital Infantil Dr. Robert Reid Cabral (Other)
Responsible Party: Principal Investigator, Justin Stoler, Asst. Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: 20140009
Record Dates: First submitted 2015-04-27; First posted 2015-05-06 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study group (Experimental): There is one group of patients which are those presenting to the hospital with suspected clinical case of dengue fever for diagnosis. This group will have oral fluid collected via the SaniSal oral fluid collector and a pipette, and blood collected via venipuncture.
  Interventions: Device: SaniSal Oral Fluid Collector

INTERVENTIONS:
Device: SaniSal Oral Fluid Collector — SaniSal is an oral fluid collector used to collect oral fluid from the mouth with an absorbant sponge.

SUMMARY:
Dengue is the most common viral illness spread by mosquitos. It is important to diagnose dengue to prompt adequate therapy and initiate local mosquito control. Easy to use point of care tests are needed to improve dengue diagnosis. Oral fluid collection may be a simple, non-invasive way to diagnose dengue in the community. However, it is currently unknown if oral fluid is an accurate way to diagnose dengue and if the use of a specialized oral fluid collector could help to improve dengue diagnosis. In this study, the investigators will analyze the oral fluid of suspected dengue patients compared to serum samples for dengue diagnosis. From this information the investigators will be able to determine if oral fluid is a convenient way to diagnose dengue and if the oral fluid collector aids in improving diagnosis.

DETAILED DESCRIPTION:
Dengue continues to spread and threaten approximately 3.6 billion people. It is crucial to adequately recognize dengue and start early intervention. Dengue virus (DENV) infections are typically confirmed by virus isolation and nucleic acid detection, both of which require trained personnel and advanced facilities that are limited in developing countries. Detection of antibodies serves as a viable and cheaper diagnostic alternative, and one method of doing so is through oral fluid. Detecting DENV antibodies in oral fluid has been accomplished. The utility of oral fluids is attractive as specimens can be acquired in a faster, non-invasive manner that is suitable for children and needle-phobic adults. One challenge of using oral fluid for dengue diagnosis is that typically, oral fluid contains the same analytes found in blood, albeit in lower concentrations, thus there is a need for protein concentration if oral fluid will be used for diagnosis.

A device capable of collecting oral fluid is the Sani-Sal® oral fluid collector, used successfully in rapid diagnostics of HIV. It is a unique device that claims to concentrate oral fluid proteins, decrease oral fluid viscosity, and stimulate salivation. These properties make the Sani-Sal® potentially valuable in the diagnosis of DENV in the field by concentrating antibodies to identify early infection.

Furthermore, dengue is commonly misdiagnosed or undiagnosed given varying clinical manifestations, lack of patient health seeking behavior, and lack of incentives for physicians to confirm and report cases. Knowledge on the health-seeking behaviors of dengue patients remains limited. The project will also assess patient and practitioner perceptions regarding dengue diagnostics, care, and reporting while considering the utility of this novel diagnostic technology. Lastly, the study will seek to understand the role of governance in communicable disease surveillance, reporting and information flow.

This application seeks approval to pilot a study which will seek to determine whether the SaniSal® can be useful in DENV diagnosis by concentrating DENV IgM antibodies and NS1 antigens. The study will also like to explore the knowledge, attitude, practices and health seeking behaviors of patients, while understanding dengue training, diagnosis and reporting amongst practitioners. The study will be conducted in partnership with the Instituto Nacional de Diabetes (INDEN) and Dr. Roberto Reid Cabral's Children's Hospital in Santo Domingo, Dominican Republic-where dengue is endemic.

The utility of oral-fluid in diagnostics is promising: it can serve as efficient tools for point-of-care practices and as an alternative to blood-draw. If this study shows that saliva can be equally effective in the detection of DENV as blood on an ELISA confirmatory test, then the investigators can mitigate the limitations of serum testing. This can result in increased rapid diagnostic confirmation of suspected cases, improving on patient comfort and care while assisting in targeted vector control. This coupled with insights on policies, perceptions and behaviors surrounding DENV can help improve point-of-care diagnostics, reporting and surveillance, and community education efforts during epidemics in endemic countries of the Caribbean region.

ELIGIBILITY:
Inclusion Criteria:

* Febrile for at least 36 hours with clinical characteristics of dengue
* Presents for care at the hospital during time of study
* Over the age of 2 years old
* Adults are able and willing to consent or a parent/guardian is willing and able to accept consent for a child.

Exclusion Criteria:

* Adults that are not able to consent
* Minors without parent/guardian consent
* Pregnant women
* Prisoners

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Dengue Immunoglobulin M (IgM) and Non-Structural Protein 1 (NS1) Concentration in Oral Fluid | up to 2 years after the beginning of the study
  IgM and NS1 Concentration via ELISA from oral fluid collected via the SaniSal Oral Fluid collector versus pipette compared to serum concentration.

SECONDARY OUTCOMES:
Patient Acceptability of Oral Fluid Collector | up to 2 years after beginning of the study
  Patient interviews about the acceptability of using an oral fluid collector for diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Justin Stoler, PhD MPH, Principal Investigator — University of Miami
Locations (1):
- Hospital Infantil, Santo Domingo, Dominican Republic

REFERENCES:
- [Background] Cabrera-Batista B, Skewes-Ramm R, Fermin CD, Garry RF. Dengue in the Dominican Republic: epidemiology for 2004. Microsc Res Tech. 2005 Nov;68(3-4):250-4. doi: 10.1002/jemt.20225. PMID 16276520
- [Background] Perez-Guerra CL, Zielinski-Gutierrez E, Vargas-Torres D, Clark GG. Community beliefs and practices about dengue in Puerto Rico. Rev Panam Salud Publica. 2009 Mar;25(3):218-26. doi: 10.1590/s1020-49892009000300005. PMID 19454149
- [Background] Parisi MR, Soldini L, Di Perri G, Tiberi S, Lazzarin A, Lillo FB. Offer of rapid testing and alternative biological samples as practical tools to implement HIV screening programs. New Microbiol. 2009 Oct;32(4):391-6. PMID 20128446
- [Background] Balmaseda A, Guzman MG, Hammond S, Robleto G, Flores C, Tellez Y, Videa E, Saborio S, Perez L, Sandoval E, Rodriguez Y, Harris E. Diagnosis of dengue virus infection by detection of specific immunoglobulin M (IgM) and IgA antibodies in serum and saliva. Clin Diagn Lab Immunol. 2003 Mar;10(2):317-22. doi: 10.1128/cdli.10.2.317-322.2003. PMID 12626461
- [Background] Yap G, Sil BK, Ng LC. Use of saliva for early dengue diagnosis. PLoS Negl Trop Dis. 2011 May 10;5(5):e1046. doi: 10.1371/journal.pntd.0001046. PMID 21572982